CLINICAL TRIAL: NCT02014259
Title: Investigation of Pharmacokinetics, Safety and Tolerability of Oral Semaglutide in Subjects With Various Degrees of Impaired Renal Function Compared to Subjects With Normal Renal Function
Brief Title: Pharmacokinetics, Safety and Tolerability of Oral Semaglutide in Subjects With Various Degrees of Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4079; 2013-000682-36 (EudraCT Number); U1111-1139-4281 (Other: WHO)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects with renal impairment (Experimental)
  Interventions: Drug: semaglutide
- Subjects with normal renal function (Active Comparator)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Once daily oral administration of semaglutide formulated with SNAC. Dose escalation, with 5 days on 5 mg followed by 5 days on 10 mg

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body), safety and tolerability of oral semaglutide in subjects with various degrees of impaired renal function compared to subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-85 years (both inclusive) at the time of signing inform consent
* Subject with normal renal function or renal impairment (mild, moderate, severe or end-stage renal disease requiring dialysis)
* For subject with normal renal function: good general health (as judged by the investigator)
* Body mass index (BMI) 18.5-40.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods
* History of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease
* Uncontrolled hypertension (defined as systolic blood pressure above or equal to 180 mmHg and/or diastolic blood pressure above or equal to 100 mmHg)
* Any blood draw or donation of blood or plasma in excess of 400 mL within the 3 months preceding the screening visit (Visit 2)
* History of significant drug abuse, or a positive drug test at the screening visit (Visit 2)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-12-11 (Actual); Primary Completion 2014-10-24 (Actual); Study Completion 2014-10-24 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration time curve | From time 0 to 24 hours after the 10th dosing

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration | 0 to 24 hours after the 10th dosing
Area under the SNAC (Sodium N-[8-(2-hydroxybenzoyl) amino] caprylate /salcaprozate sodium) plasma concentration time curve | From time 0 to 24 hours after the 10th dosing
Maximum observed SNAC plasma concentration | 0 to 24 hours after the 10th dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Czechia (2):
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Prague
- Novo Nordisk Investigational Site, Budapest, Hungary

REFERENCES:
- [Result] Granhall C, Sondergaard FL, Thomsen M, Anderson TW. Pharmacokinetics, Safety and Tolerability of Oral Semaglutide in Subjects with Renal Impairment. Clin Pharmacokinet. 2018 Dec;57(12):1571-1580. doi: 10.1007/s40262-018-0649-2. PMID 29623579
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com